CLINICAL TRIAL: NCT03823573
Title: Prospective Clinical Trial Regarding the Implementation of a Rapid Recovery Protocol in Total Knee Arthroplasty in Rio Hortega University Hospital
Brief Title: Implementation of a Rapid Recovery Protocol in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ignacio Aguado Maestro (Other)
Responsible Party: Sponsor-Investigator, Ignacio Aguado Maestro, Principal Investigator, Hospital del Rio Hortega
Organization: Hospital del Rio Hortega (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: P1102-16
Record Dates: First submitted 2019-01-27; First posted 2019-01-30 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Fast Track; Tranexamic Acid Adverse Reaction; Knee Osteoarthritis
Keywords: fast track; total knee arthroplasty; tranexamic acid; drain
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Drainage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid recovery protocol (Experimental): They will start walking the day of surgery. Levobupivacain 5mg/ml will be placed in the knee tissues. Tranexamic acid inside the knee. No drains.
  Interventions: Behavioral: Walk within 24 hours
- Classic protocol (Active Comparator): They will start walking 3 days after surgery. Levobupivacain 5 mg/ml will be placed in the femoral nerve. Tranexamic acid inside the knee. A Redon drain will be used.
  Interventions: Behavioral: Walk within 24 hours

INTERVENTIONS:
Behavioral: Walk within 24 hours — Patients will start walking on different timings. Patients on the rapid recovery protocol won't be using drains.
  Other Names: Drain; Discharge the day after walking

SUMMARY:
Patients undergoing total knee arthroplasty will follow two different rehabilitation protocols. In one of them, they will start walking the day of surgery and discharged on a 48 hours basis. On the other one, start walking 3 days after surgery and discharged on a 96 hours basis. Outcomes will be satisfaction, pain, range of movement, incidence of DVT and overall complications.

DETAILED DESCRIPTION:
Randomization will be performed concealed the day before surgery. Tranexamic acid will be used in both groups. Rapid recovery group will not be using a drain, whereas the standard protocol group will have one.

ELIGIBILITY:
Inclusion Criteria:

* Knee osteoarthritis willing to undergo total knee arthroplasty
* Age 55-79
* Consent

Exclusion Criteria:

* Hipersensibility to any of the components used
* Epilepsy
* Pulmonary embolism

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Pain: Morphine clorhydrate shots requested by the patient | 24 hours
  Number of shots requested and administered to the patient after surgery
Range of Motion | 6 months
  Knee range of motion measured in degrees of flexion (0-180º and extension (0-180º)
Ultrasonography incidence of deep vein thrombosis | 4 weeks-8 weeks
  Incidence of deep vein thrombosis measured by ultrasound
Overall score given by the patient to the knee replacement process | 6 months
  Satisfaction with the protocol. Subjective measure by the patient from 0 (bad) to 10 (best) with the surgery process.
Infection | 1 year
  Incidence of infection
Blood loss | 48 hours
  Haemoglobin drop
Oxford Knee Score pre op and post op | 6 months
  Difference in Oxford Knee Scores postoperatively and preoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario del Río Hortega, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No